CLINICAL TRIAL: NCT04008004
Title: A Phase 1a/1b Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of EDP 514 in Healthy Subjects (Part 1), and Antiviral Activity in Nucleos(t)Ide Reverse Transcriptase Inhibitor (NUC)-Suppressed Patients With Chronic Hepatitis B Virus Infection (Part 2)
Brief Title: A Study of EDP-514 in Healthy Subjects (Part 1) and Patients With Chronic Hepatitis B Virus Infection (Part 2)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Collaborators: Pharmaceutical Research Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EDP 514-001
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-05

CONDITIONS: Chronic HBV Infection
Keywords: "First-in-Human"; Single Ascending Dose; Multiple Ascending Dose; hepatitis B virus; HBV
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- EDP-514 HV SAD Cohorts (Experimental): EDP-514 Dose 1, Dose 2, Dose 3, Dose 4, Dose 5 and Dose 6 orally, once daily in one single administration
  Interventions: Drug: EDP-514
- EDP-514 HV MAD Cohorts (Experimental): EDP-514 Dose 1, Dose 2 and Dose 3 orally, once daily for 14 days
  Interventions: Drug: EDP-514
- EDP-514 HV SAD Placebo Cohort (Placebo Comparator): Matching placebo, orally, once daily in one single administration
  Interventions: Drug: Placebo
- EDP-514 HV MAD Placebo Cohort (Placebo Comparator): Matching placebo, orally, once daily for 14 days
  Interventions: Drug: Placebo
- EDP-514 HBV MAD Cohorts (Experimental): EDP-514 Dose 1, Dose 2 and Dose 3 orally, once daily for 28 days
  Interventions: Drug: EDP-514
- EDP-514 HBV MAD Placebo Cohort (Placebo Comparator): Matching placebo, orally, once daily for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP-514 — Oral Capsule; Subjects will receive either a single dose of EDP-514 on Day 1 only (SAD HV), once daily dosing of EDP-514 starting on Day 1 through Day 14 (MAD HV) or once daily dosing of EDP-514 starting on Day 1 through Day 28 (MAD HBV).
  Arms: EDP-514 HBV MAD Cohorts; EDP-514 HV MAD Cohorts; EDP-514 HV SAD Cohorts
Drug: Placebo — Placebo to match EDP-514
  Arms: EDP-514 HBV MAD Placebo Cohort; EDP-514 HV MAD Placebo Cohort; EDP-514 HV SAD Placebo Cohort

SUMMARY:
Part 1 is a randomized, double-blind, placebo-controlled study. It will assess the safety, tolerability, and pharmacokinetics of single and multiple orally administered doses of EDP-514 in healthy adult subjects.

Part 2 is randomized, double -blind, placebo-controlled study including subjects with Hepatitis B Virus. It will assess the safety, tolerability, pharmacokinetics and antiviral activity of 28 Days of orally administered doses of EDP-514 in nucleos(t)ide reverse transcriptase inhibitor (NUC)-Suppressed Patients with Chronic Hepatitis B Virus Infection

DETAILED DESCRIPTION:
Part 1 consists of two phases planned in healthy subjects:

The first phase assesses single ascending doses for EDP-514 (active drug or placebo) in healthy subjects. A "fasted" and "fed" two-part cohort will also assess food effect.

The second phase assesses multiple ascending doses (active drug or placebo) for 14 days in healthy subjects.

Each cohort within each phase will enroll a total of 8 subjects who will be randomized to receive EDP-514 or placebo. The cohort assessing food effect will enroll 10 subjects randomized to receive EDP-514 or placebo.

Part 2 assesses multiple ascending doses EDP-514 (active drug or placebo) for 28 days in nucleos(t)ide reverse transcriptase inhibitor (NUC)-Suppressed Patients with Chronic Hepatitis B Virus Infection.

Each cohort in Part 2 will enroll a total of 8 subjects who will be randomized to receive EDP-514 or placebo.

ELIGIBILITY:
Part 1 (HV Population):

Inclusion Criteria:

* An informed consent document signed and dated by the subject.
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 65 years, inclusive.

Exclusion Criteria:

* Clinically relevant evidence or history of illness or disease.
* Pregnant or nursing females.
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection.
* A positive urine drug screen at screening or Day -1.
* Current tobacco smokers or use of tobacco within 3 months prior to screening.
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy).
* History of regular alcohol consumption.
* Receipt of any vaccine, an investigational agent or biological product within 28 days or 5 times the t½, whichever one is longer, prior to first dose. This includes agents administered during clinical trial participation.

Part 2 (HBV Population):

Inclusion Criteria:

* An informed consent document signed and dated by the subject.
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 70 years, inclusive
* HBV DNA levels:

  * A Screening HBV DNA level in serum/plasma that is <LLOQ and
  * No HBV DNA serum/plasma test values ≥LLOQ over the previous 12 months (using an approved test)
* CHB subjects must have been on their prescribed HBV NUC treatment with no change in regimen for 12 months prior to Screening

Exclusion Criteria:

* A documented prior diagnosis of cirrhosis
* Pregnant or nursing females
* Coinfection with human immunodeficiency virus (HIV), HCV, HDV, HAV, or HEV
* Chronic liver disease of a non-HBV etiology; coexisting liver or biliary diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Safety measured by adverse events | Up to 8 Days in HV SAD Cohorts
Safety measured by adverse events | Up to 21 Days in HV MAD Cohorts
Safety measured by adverse events | Up to 56 Days in HBV MAD Cohorts

SECONDARY OUTCOMES:
Cmax of EDP-514 | Up to 6 Days in HV SAD Cohorts
AUC of EDP-514 | Up to 6 Days in HV SAD Cohorts
Cmax of EDP-514 | Up to 18 Days in HV MAD Cohorts
AUC of EDP-514 | Up to 18 Days in HV MAD Cohorts
Cmax of EDP-514 | Up to 28 Days in HBV MAD Cohorts
AUC of EDP-514 | Up to 28 Days in HBV MAD Cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (15):
- United States (11):
  - Southern California GI and Liver Centers, Coronado, California
  - University of California Los Angeles, Los Angeles, California
  - Tuan Nguyen Md Gastroenterology & Hepatology (Tuan Nguyen, M.D., Inc.), San Diego, California
  - Quest Clinical Research, San Francisco, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - Pharmaceutical Research Associates, Inc., Lenexa, Kansas
  - Digestive Disease Associates - Catonsville, Catonsville, Maryland
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - American Research Corporation, Houston, Texas
  - The Texas Liver Institute, San Antonio, Texas
  - Swedish Organ Transplant and Liver Center, Seattle, Washington
- Canada (4):
  - University Of Calgary, Calgary, Alberta
  - Gastroenterology Institute of Research Institute, Vancouver, British Columbia
  - Toronto General Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec